CLINICAL TRIAL: NCT04229485
Title: The Chinese Cohort Study of Chronic Kidney Disease Patients Followed on Smartphone Platform, a Multi-center Observational Study
Brief Title: Chinese Chronic Renal Insufficiency Study: Based on Smartphone Platform
Acronym: C-CRISS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Limeng Chen (Other)
Collaborators: First Hospital of China Medical University (Other); People's Hospital of Xinjiang Autonomous Region (Unknown); Fujian Provincial Hospital (Other); Qianfoshan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); People's Hospital of Ningxia Hui Autonomous Region (Other)
Responsible Party: Sponsor-Investigator, Limeng Chen, Professor of Medicine, Associate Chief of Nephrology Division, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: C-CRISS
Record Dates: First submitted 2019-12-29; First posted 2020-01-18 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney diseae; mineral bone disease; cardiovascular events; mobile communication
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, 24 hour urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center prospective cohort study. The purpose of this study is to investigate the relationship between bone metabolic markers and other non-traditional risk factors with kidney function progression, cardiovascular and cerebrovascular diseases, and bone loss in patients with CKD G3-5ND. In the meantime, this study is to explore a new mode of management and complication monitoring through mobile communication in chronic kidney disease patients.

DETAILED DESCRIPTION:
Abnormal mineral bone metabolism of chronic kidney disease (CKD-MBD) is the most common complication of CKD. It involves kidney, bone metabolism, parathyroid gland, cardiovascular and cerebrovascular organs. It is an independent risk factor for progression of CKD to end-stage renal disease (ESRD), vascular and cardiac valve calcification, and cardiovascular and cerebrovascular events. However, less data concerning the relationship between bone metabolic index, such as high blood phosphorus and cardiovascular diseases, bone mass reduction and fracture is available in Chinese adult patients. This study is a multi-center prospective cohort study to explore the relationship between bone metabolic markers and other non-traditional risk factors with renal function progression, cardiovascular and cerebrovascular diseases, and bone loss in patients with CKD G3-5ND. Based on the sample size estimation, 3360 subjects should be enrolled in this study. The primary outcome is progression to ESRD (start dialysis or kidney transplantation) or doubling of serum creatinine, as well as cardiovascular events and all-cause mortality.

At present, the follow-up and the management of complications of CKD patients are not enough. The popularity of mobile communication in China provide the possibility to strengthen the follow-up and complications management in CKD patients and save human resources. This study is to explore a new mode of collecting datas through mobile communication in chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

* at least two measurements of serum Cr (with a minimum interval of 3 months), , 10≤eGFR≤60ml/min/1.73m^2

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Patients attending oncology, psychiatry, human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS), viral hepatitis (HBV or HCV) services
* Acute mycardial infarction within the last six months
* NYHA Class III or IV heart failure at baseline
* Ongoing chemotherapy or immunosuppressive therapy (in the preceding 6 months to treat renal or immune disease)
* Current renal replacement therapy
* Current pregnancy or breastfeeding women
* Any organ transplantation
* Currently participation in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients stage 3-5ND
Sampling Method: Non-Probability Sample
Enrollment: 3360 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of progression to ESRD | 2 year
  begin to dialysis and kidney transplantation
cardiovascular event and all-cause mortality | 2 year
  diagnose as myocardial infarction, heart failure, stroke and cerebral hemorrhage

SECONDARY OUTCOMES:
the rate of eGFR decline | 2 years
  the rate of eGFR decline
bone mass change | 2 years
  the bone mass change based on DXR
Kidney Disease Outcomes Quality Initiative-Short Form 36 | 2 years
  the scores change of Kidney Disease Outcomes Quality Initiative- Short Form 36 The score of Kidney Disease Outcomes Quality Initiative-Short Form 36 is between 0 and 100. The higher score means a better self-evaluation.
frailty | 2 years
  A frailty phenotype was established with five variables: unintentional weight loss, self-reported exhaustion, low energy expenditure, weak grip strength and low gait speed. Those with three or more of the five factors were judged to be frail, those with one or two factors as pre-frail, and those with no factors as not frail.
the way of dialysis initiation | 2 years
  record if the patient start dialysis with urgency and mode of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, MD, PhD, Principal Investigator — Division of Nephrology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To comply with laws in China, local regulations and hospital policy, IPD sharing might be restricted

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] Bello AK, Alrukhaimi M, Ashuntantang GE, Basnet S, Rotter RC, Douthat WG, Kazancioglu R, Kottgen A, Nangaku M, Powe NR, White SL, Wheeler DC, Moe O. Complications of chronic kidney disease: current state, knowledge gaps, and strategy for action. Kidney Int Suppl (2011). 2017 Oct;7(2):122-129. doi: 10.1016/j.kisu.2017.07.007. Epub 2017 Sep 20. PMID 30675426
- [Background] Dienemann T, Fujii N, Orlandi P, Nessel L, Furth SL, Hoy WE, Matsuo S, Mayer G, Methven S, Schaefer F, Schaeffner ES, Sola L, Stengel B, Wanner C, Zhang L, Levin A, Eckardt KU, Feldman HI. International Network of Chronic Kidney Disease cohort studies (iNET-CKD): a global network of chronic kidney disease cohorts. BMC Nephrol. 2016 Sep 2;17(1):121. doi: 10.1186/s12882-016-0335-2. PMID 27590182
- [Background] Zhou C, Wang F, Wang JW, Zhang LX, Zhao MH. Mineral and Bone Disorder and Its Association with Cardiovascular Parameters in Chinese Patients with Chronic Kidney Disease. Chin Med J (Engl). 2016 Oct 5;129(19):2275-80. doi: 10.4103/0366-6999.190678. PMID 27647184